CLINICAL TRIAL: NCT00722241
Title: Effectiveness and Safety Study of the Next-Generation DexCom™ SEVEN® Continuous Glucose Monitoring System
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Andrew K. Balo / SVP, Clinical and Regulatory Affairs, and Quality Assurance, DexCom, Inc.
Other Study IDs: PTL-300012, Rev01
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Continuous Glucose Monitoring; Interstitial Fluid; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Adult subjects (at least 18 years of age) with a diagnosis of type 1 diabetes (~80%) or insulin-treated type 2 diabetes (~20%); method of insulin delivery may be multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the next-generation DexCom SEVEN Continuous Glucose Monitoring System (SEVEN.2 System) when worn for up to 7-days by subjects >18 years-old with diabetes mellitus requiring insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Have been diagnosed with insulin-requiring diabetes and are on multiple daily injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII) insulin therapy
* Willing not to inject insulin or wear an insulin pump insertion set within 3 inches from the Sensor site during Sensor wear
* Willing to use only the blood glucose meter(s) provided to them for self-monitoring of blood glucose (SMBG) during Sensor wear
* Willing to participate in one, 8-hour in-clinic session and be willing to take 4 fingersticks per hour and have 4 blood draws per hour for the entire 8-hour duration
* Willing to take a minimum of 6 fingersticks per day during home use (2 for calibration purposes, 4 for comparative purposes)
* Willing to refrain from the use of acetaminophen during the Sensor insertion period and for at least 24-hours prior to Sensor insertion
* Willing not to schedule a magnetic resonance (MRI) scan, computed tomography (CT) scan, or x-ray, for the duration of the study
* Able to speak, read, and write English

Exclusion Criteria:

* Have extensive skin changes/diseases that preclude wearing the Sensor on normal skin (e.g. extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites
* Subjects who have a known allergy to medical-grade adhesives
* Are pregnant as demonstrated by a positive pregnancy test within 72 hours of insertion
* Have a hematocrit that is less than 30%, or greater than 55%
* Current participation in another investigational study protocol (if a subject has recently completed participation in another drug study, the subject must have completed that study at least 30 days prior to being enrolled in this study)
* Have any condition that, in the opinion of the Investigator, would interfere with their participation in the trial or pose an excessive risk to study staff handling venous blood samples (e.g., known history of hepatitis B or C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory (non-hospitalized) individuals with type 1 diabetes or insulin-treated type 2 diabetes selected from endocrinology clinics within the United States
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
SEVEN.2 System accuracy as compared to Yellow Springs Instrument (YSI) venous blood glucose measurements | Days 1, 4, and 7 of Sensor wear

CONTACTS AND LOCATIONS:
Overall Officials: Andrew K Balo, BS, Study Chair — DexCom, Inc.
Locations (3):
- United States (3):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Advanced Metabolic Care + Research, Escondido, California
  - Sansum Diabetes Research Institute, Santa Barbara, California